CLINICAL TRIAL: NCT02234674
Title: Pilot Efficacy Study of the Stendo Pulsating Suit in Patient With Leg Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stendo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00355-42
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2014-09

CONDITIONS: Primary Lower Limb Lymphedema; Secondary Lower Limb Lymphedema
Keywords: Pulsating suit; lymphedema; leg volume
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard intensive CDP (Active Comparator): This arm is the controlled group ; patients in that group will undergo a current practice performed in the lymphology unit.
  Interventions: Other: Current intensive CDP
- Stendo group (Experimental): This arm contitutes the group where the Stendo pulsating suit sessions are investigated in the frame of the CDP in replacement of the pressotherapy sessions.
  Interventions: Other: intensive CDP where Stendo pulsating suit replaces pressotherapy

INTERVENTIONS:
Other: Current intensive CDP — Standard Intensive CDP including
  * manual lymph drainage,
  * pressotherapy and
  * bandaging
  Arms: Standard intensive CDP
Other: intensive CDP where Stendo pulsating suit replaces pressotherapy — The intervention consist to perform daily during 5 days an intensive CDP where pressotheray is replaced by Stndo pulsating suit sessions.
  Arms: Stendo group

SUMMARY:
This study aims at evaluating the efficacy of the Stendo pulsating suit in patients with a leg lymphedema hospitalized for intensive Complex Decongestive Physiotherapy (CDP).

This study is a pilot controlled randomized study with two arms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a primary or secondary lympedema clinically diagnosed (Stemmer Sign) of one or two legs.
* Patient with a lympedema stage II (persistent) or III according to the classification of the International Society of Lymphoedema (ISL)
* Patient aged 18 or more

Exclusion Criteria:

* Patient with a severe heart, kidney or liver failure,
* Patient with an advanced obstructive arterial disease
* Patient with a recent and progressive deep venous thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
volume of the most affected leg | baseline ; after 5 days intensive CDP
  Change in % of the volume of the most affected leg according to disk model method

SECONDARY OUTCOMES:
Quality of Life | baseline ; after 5 days intensive CDP
  36 health survey questionnaire (SF-36) and Visual Analogical Scale

CONTACTS AND LOCATIONS:
Locations (1):
- CHIC Des Andaines, La Ferté-Macé, France

REFERENCES:
- [Result] Deltombe T, Jamart J, Recloux S, Legrand C, Vandenbroeck N, Theys S, Hanson P. Reliability and limits of agreement of circumferential, water displacement, and optoelectronic volumetry in the measurement of upper limb lymphedema. Lymphology. 2007 Mar;40(1):26-34. PMID 17539462
- [Result] Mayrovitz HN, Macdonald J, Davey S, Olson K, Washington E. Measurement decisions for clinical assessment of limb volume changes in patients with bilateral and unilateral limb edema. Phys Ther. 2007 Oct;87(10):1362-8. doi: 10.2522/ptj.20060382. Epub 2007 Aug 7. PMID 17684090